CLINICAL TRIAL: NCT05452382
Title: Surgical Outcome and Predictors of Overall Survival of Stage I-III Appendiceal Adenocarcinoma; a National Cancer Database Analysis
Brief Title: Surgical Outcome and Predictors of Overall Survival of Stage I-III Appendiceal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Collaborators: Cleveland Clinic Florida (Other)
Responsible Party: Principal Investigator, Sameh Emile, Research associate, Cleveland Clinic Florida
Other Study IDs: NCDBAppendix
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Appendiceal Cancer
MeSH Terms: conditions — Appendiceal Neoplasms | interventions — Colectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Partial colectomy: Patients with appendiceal cancer who underwent segmental resection of appendiceal adenocarcinoma
  Interventions: Procedure: Partial colecctomy
- Hemicolectomy: Patients with appendiceal cancer who underwent formal right hemicolectomy of appendiceal adenocarcinoma
  Interventions: Procedure: Hemicolectomy

INTERVENTIONS:
Procedure: Partial colecctomy — Segmental resection of appendiceal adenocarcinoma including terminal ileum and cecum
  Groups: Partial colectomy
Procedure: Hemicolectomy — Formal right hemicolectomy including terminal ileum, cecum, and ascending colon
  Groups: Hemicolectomy

SUMMARY:
A few studies investigated the predictors of overall survival in appendiceal adenocarcinoma. A SEER database analysis of 1404 patients with appendiceal adenocarcinoma found that older age, T4 tumors, N1-2 stage, poorly differentiated carcinoma, and distant metastasis were significantly predictive of poorer survival. Another small single-center study including 49 appendiceal cancer patients reported female gender and low-grade adenocarcinoma to be associated with increased overall survival. However, these previous analyses did not take into account some important prognosticators of survival such as patients' comorbidities and functional status, pathologic parameters such as lymphovascular invasion, and adjuvant systemic treatment. Therefore, we used the National Cancer Database (NCDB) to conduct a comprehensive analysis of the predictors of overall survival after surgical treatment of stage I-III appendiceal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-metastatic appendiceal adenocarcinoma who underwent surgical resection

Exclusion Criteria:

* Patients with other pathologic types of appendiceal cancer
* Patients with clinical stage IV or unknown stage
* Patients who did not undergo surgery, underwent local excision, or had unknown/non-specified surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with stage I-III appendiceal adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 2607 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-07-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 60 months
  Percent of patients who were alive at five years of follow-up

SECONDARY OUTCOMES:
Positive resection margins | Immediate postoperative
  the rate of surgical margins infiltrated by malignancy

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic Flroida, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: No